CLINICAL TRIAL: NCT06633484
Title: BIOmarkers of MIGraine: a Proof of Concept Study on the Stratification of Responders to CGRP Monoclonal Antibodies - Results from Magnetic Resonance Imaging
Brief Title: BIOMIGA: Results from Magnetic Resonance Imaging
Status: Active, not recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMIGA-MR
Record Dates: First submitted 2024-07-30; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Migraine
Keywords: brain morphology; neuronal functional connectivity; CGRP-Antibodies
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Migraine patients
  Interventions: Other: functional magnetic resonance imaging
- Healthy Controls
  Interventions: Other: functional magnetic resonance imaging

INTERVENTIONS:
Other: functional magnetic resonance imaging — non-diagnostic, non-invasive, passive measurement of the brain's structure and function

SUMMARY:
The projects comprising in the multicenter BIOMIGA project have been preregistered earlier with ID NTC04503083 at clinicaltrials.gov. Here the imaging subproject within the overall BIOMIGA aims is specified. The hypotheses for this subproject of the magnetic resonance imaging part is based on hypotheses generating analyses of the data from one site (Hamburg, Germany) of this three-center study. At all three sites healthy controls and migraine patients underwent identical protocols with 3 types of magnetic resonance imaging including structural scans (MPRAGE), resting-state functional magnetic resonance imaging (rs-fMRI) as well as arterial spin labeling (ASL) with matched protocols across sites. Data was acquired before CGRP-antibody administration (day 1) and 12 weeks afterwards (day 2). We analyzed the data from one site (Hamburg, Germany) as hypotheses generating, published these data as a poster and aim to validate our results with the not-yet analyzed data from the two other sites (Pavia, Italy and Barcelona, Spain).

DETAILED DESCRIPTION:
The Hamburg data was processed as stated below and will be used as independent data set for hypotheses generation. The data of the two other sites (Italy and Spain) will be processed identically to the Hamburg data set:

rs-FMRI

Preprocessing of the resting-state functional MR data followed the SPM12 pipeline (https://www.fil.ion.ucl.ac.uk/spm/software/spm12/) using slice time correction, realignment, coregistration to the structural image, normalization into MNI space, and smoothing with an 8mm^3 Gausian kernel. Data was further analyzed using the CONN-toolbox (https://web.conn-toolbox.org/) where a 0.003-0.08 Hz temporal filter and denoising with linear regression of confounding effects (white matter, CSF, movement) and linear detrending. We choose:

* Local Homogeneity (LCOR),
* Global Correlations (GCOR),
* Seed-Based Correlations (SBC): Seed to voxel and ROI to ROI with an additional mask of the hypothalamus
* Independent Component Analyses (group-ICA),
* Amplitude of Low-Frequency Fluctuations (ALFF)

Statistical comparisons calculated are defined as primary and secondary outcomes below and include (i) prediction of treatment outcome (reduction in headache days) from T0 (further PR), (ii) alterations between T0 and T1, (iii) differences between healthy controls and migraine patients at T0 (further HvsPAT), and (iv) differences between responders and non-responder at T0 and T1.

In the hypothesis generating Hamburg data significant results at a threshold of cluster-wise FDR-corrected p<0.05 with an entry threshold of voxel-wise uncorrected p<0.001, when corrected for age and sex in were found:

* LCOR: PR: Two clusters in left lateral occipital cortex and right temporal fusiform cortex; HvsPAT: bilateral thalamus left frontal operculum.
* SBC Seed to Voxel: PR: Hypothalamus 2 clusters, Sensori Motor Lateral R 1 cluster, Visula Lateral L 1 cluster, Visual Lateral R 3 cluster; HvsPAT: Sensori Motor Lateral L 5 cluster, Sensori Motor Lateral R 1 cluster, Sensori Motor Superior 3 cluster, Visual Medial 3 cluster, Visual Occipital 1 cluster, Visual Lateral L 4 cluster, Visual Lateral R 1 cluster,
* ICA: ICA 5 2 cluster, ICA 16 2 cluster, ICA 28 1 cluster, ICA 34 2 cluster; HvsPAT: ICA 4 3cluster, ICA 6 4 cluster, ICA 14 4 cluster, ICA 18 2 cluster, ICA 27 3 cluster, ICA 29 14 cluster, ICA 33 3 cluster, ICA 36 7 cluster, ICA 38 6 cluster
* There were no significant results for SBC ROI to ROI, GCOR and ALFF
* There were no significant results for the chosen threshold for the comparisons between responders and non-responder at T0 and T1 Preliminary results for local and global connectivity were recently presented at a scientific conference.

To reproduce the significant results from the Hamburg data there is choosen a small volume-corrected threshold of p<0.05. For non-significant result, the statistical threshold for the data of the two other sites will be set to voxel-wise FWE-corrected p<0.05.

MPRAGE Raw T1-images (aka MPRAGE) were processed using the CAT12-toolbox (https://neuro-jena.github.io/cat12-help/) which extents SPM12 (https://www.fil.ion.ucl.ac.uk/spm/software/spm12/). For controls and migraine patients with data from only the first day, images segmented into compartments of gray and white matter and normalized. For patients with data from 2 days, data was longitudinally segmented. Images of gray and white matter were smoothed with an isotropic Gaussian kernel of 6 mm3. T-test and F-tests implemented in the SPM12 toolbox were used to estimate significant differences at a threshold of cluster-wise-correct p<0.05. The individual total intracranial volume (TIV), which is also estimated by the CAT12-toolbox, was used as covariate to control for different brain sizes. Age and gender were used as further covariates when indicated. All results were masked by gray or white matter masks stemming from a segmentation of the average normalized T1s of the participants. The statistical threshold for the hypotheses generating data set from Hamburg was set to cluster-wise FDR-corrected p<0.05 with an entry threshold of voxel-wise uncorrected p<0.001. As no significant results were achieved, the statistical threshold for the data of the two other sites will be set to voxel-wise FWE-corrected p<0.05.

ASL ASL was not yet analyzed for any of the sites. For the statistics we will use Cerebral Perfusion Images stemming from the toolbox ASLtbx (https://www.cfn.upenn.edu/zewang/ASLtbx_manual.pdf). Nevertheless, as different imaging protocols were available in Spain and Italy, a comparison of the equality has to be proofen first. Therefore, we acquired both protocols in the Hamburg data. As we do not expect any differences here, the statistical threshold will be set to voxel-wise FWE-corrected p<0.05.

Power calculation based on Hamburg MR data Power analysis of the primary outcome "prediction of headache reduction with resting-state functional connectivity measures from fMRI of day 1" for which rs-fMRI data of 54 migraine patients from the hypothesis generating site Hamburg were analyzed using the CONN-toolbox revealed that 37 migraine patients are necessary to reproduce the result of significant comodulation in local correlation when corrected for age and gender (80% Power, FWE-corrected p<0.05 calculated with PowerMap). Initial quality checks of the data from the other two sites reveal enough available data for reproduction.

ELIGIBILITY:
Inclusion Criteria:

Migraine patients

* Adults between 25 and 55 years of age of both sexes;
* Patients diagnosed with high-frequency migraine (HFM) 8 or more migraine days/month) or CM with or without aura (>15 headache days migraine/month, of which 8 have migraine characteristics) according to the International Classification of Headache Disorders, 3rd edition, (ICHD-3);
* Females had to be postmenopausal for at least one year, surgically sterile or otherwise incapable of pregnancy, or using an acceptable method of birth control.

Healthy controls

* Adults between 25 and 55 years of age of both sex;
* Absence of any past, or first-degree familial history of recurrent primary or secondary headache disorders.

Exclusion Criteria:

For the clinical population:

* Headache on more than 25 days/month in the last 3 months;
* Medication overuse according to the ICHD-3 criteria.

For the entire study population (migraine and healthy controls)

* Presence of any other significant medical condition (neurological disorders, severe psychiatric illness or cardiovascular disease);
* Evidence of drug, smoking or alcohol abuse or dependence within 12 months prior to V1, based on medical records or patient self-report. An alcohol consumption >100g/week will be considered as an abuse;
* Pregnant or breastfeeding women;
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant who are not on contraception;
* Concomitant use of other migraine preventive drugs that may interfere with the endpoints of the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Migraine patients and Healthy controls. The healthy controls where recruited among hospital staff and non-related acquaintances of the patients. All migraine patients enrolled in the study have been treated with CGRP-targeting mABs according to the indications approved by the respective National regulatory bodies(Germany, Spain, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 219 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
resting state fMRI | 1 year
  Prediction of reduction in number of headache days at day 1. The statistical threshold will will be set to a small-volume corrected p<0.05 in the combined data from Barcelona and Pavia.
Morphological MR | 1 year
  Prediction of reduction in number of headache days by gray and white matter density at day 1. The statistical threshold for the data of the two other sites will be set to voxel-wise FWE-corrected p<0.05.
Arterial Spin Labelling MR | 1 year
  Prediction of reduction in number of headache days by brain perfusion at day 1. ASL was not yet analyzed for any of the sites. For the statistics we will use Cerebral Perfusion Images stemming from the toolbox ASLtbx (https://www.cfn.upenn.edu/zewang/ASLtbx_manual.pdf). The statistical threshold will be set to voxel-wise FWE-corrected p<0.05.

SECONDARY OUTCOMES:
resting-state fMRI | 1 year
  Comparison of responders and non-responders differences in rs-fMRI functional connectivity, morphometry and perfusion changes at day1. The statistical threshold for the data of the two other sites will be set to voxel-wise FWE-corrected p<0.05.
Morphological MRI, resting-state fMRI and arterial spin labelling MRI | 1 year
  Comparison of rs-fMRI functional connectivity, morphometry and perfusion changes from day1 and day2. The statistical threshold will be set to voxel-wise FWE corrected p<0.05.
Morphological MRI, resting-state fMRI and arterial spin labelling MRI | 1 year
  Comparison of rs-fMRI functional connectivity, morphometry and perfusion changes between healthy controls and migraine patients at day1. Significance will be set to a small-volume corrected threshold of p<0.05 in the combined data from Barcelona and Pavia.

CONTACTS AND LOCATIONS:
Locations (3):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- IRCCS Mondino Foundation, Pavia, Italy
- Vall d'Hebron Institute of Research, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hougaard A, Gaist D, Garde E, Iversen P, Madsen CG, Kyvik KO, Ashina M, Siebner HR, Madsen KH. Lack of reproducibility of resting-state functional MRI findings in migraine with aura. Cephalalgia. 2023 Nov;43(11):3331024231212574. doi: 10.1177/03331024231212574. PMID 37950678
- [Background] Schönthaler, M.G.F., Basedau, H., May, A., Mehnert, J., 2024. Connectivity within the visual cortex predicts the efficacy of CGRP antibodies in migraine patients. DGKN 2024, Frankfurt, Germany and Clinical Neurophysiology 159, e22
- See also: SPM12: Toolbox for preprocessing of (f)MRI data — https://www.fil.ion.ucl.ac.uk/spm/software/spm12/
- See also: CONN: Toolbox for analysis of resting-state fMRI data — https://web.conn-toolbox.org/
- See also: CAT12: Toolbox for analysis of structural MRI data (MPRAGE/T1) — https://neuro-jena.github.io/cat12-help/
- See also: ASLtbx: Toolbox for analysis of aterial-spin-labellingMRI data — https://www.cfn.upenn.edu/zewang/ASLtbx_manual.pdf